CLINICAL TRIAL: NCT04707443
Title: Correlation Between Enteral Nutrition and Early Prognosis in Infants Aged Under 6 Months Following Enterostomy
Brief Title: Enteral Nutrition in Infants With Ileostomy
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Qian Tian, Deputy Director of clinical Nutrition, Children's Hospital of Fudan University
Other Study IDs: (2020)288
Record Dates: First submitted 2020-12-31; First posted 2021-01-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Nutrition of Ileostomy Infants
Keywords: ileostomy; Human breast milk; Enteral nutrition; extensive hydrolyzed formula; amino acid formula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- enteral nutrition: Infants, undergo enterostomy for various reasons within the age range of 0-6 months.The enteral nutrition can be administered orally or via enteral nutrition, including breast milk, preterm formula, infant formula, extensive hydrolyzed formula or amino acid formula et al .To observe and study the efficacy, safety and tolerance of enteral nutrition in infants after enterostomy.

SUMMARY:
This study is a prospective, single center, practical, and observational open clinical study.

DETAILED DESCRIPTION:
Infant enterostomy is one of the emergency surgeries in pediatric gastroenterology. The most common underlying conditions during infancy include necrotizing enterocolitis, intestinal necrosis, intestinal perforation, and congenital gastrointestinal malformations. Necrotizing enterocolitis also serves as a major cause of short bowel syndrome in infants. Infants with small bowel stoma leading to short bowel syndrome face a higher incidence of complications compared to adults. Additionally, small intestinal stomy inevitably come with various complications such as infection, electrolyte imbalance, nutrient deficiencies, and malnutrition.

Currently, both domestic and international studies have shown that breast milk is the preferred choice for infant nutrition. The benefits of breastfeeding have been widely reported. For postoperative infants with digestive tract surgery, breast milk's immunoglobulins and prebiotics can help promote beneficial gut bacteria and bioactive proteins (such as lactoferrin, lysozyme, and lipoproteins), growth factors that facilitate intestinal adaptation and maturation processes while enhancing feeding tolerance and preventing infections or inflammatory disorders.

However, according to literature reports on clinical practice operations after digestive tract surgery even if early breastfeeding was initiated in 88% of cases; only 44% of infants were still being breastfed at discharge. This is due to feeding intolerance following breastfeeding which manifests as gastric retention, abdominal distension, diarrhea etc., not only delaying growth but also prolonging hospital stay while causing other adverse clinical outcomes. Some discharged infants who started breastfeeding experienced diarrhea and dehydration leading to readmission. Clinically speaking this issue has often been addressed by substituting feeds with enteral nutrition preparations (deep hydrolyzed formulas or free amino acid formulas).

The objective of this study is to assess the impact of enteral nutrition, which involves selecting appropriate preparations and human breast milk based on the child's intestinal tolerance, on growth and developmental outcomes in children following enterostomy. Additionally, we aim to investigate its effects on postoperative intestinal permeability, stoma output, gut microbiota and metabolites, sepsis incidence, colitis occurrence as well as bile stasis.

ELIGIBILITY:
Inclusion Criteria:

* After birth, infants aged 0-6 months (including neonates) undergo small bowel ostomy for various reasons.

Exclusion Criteria:

* Primary liver and kidney dysfunction, congenital multiple malformations and chromosomal abnormalities.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants, undergo enterostomy for various reasons within the age range of 0-6 months
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2021-07-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Z-scores of body weight | 4 weeks after enteral feeding
  The patient will be weighed in the recumbent position on an electronic infant scale. Z-scores for weight for age (WAZ) was obtained from the World Health Organization Anthro software and WHO Child Growth Standards.

SECONDARY OUTCOMES:
Z-scores of body length | 4 weeks day after enteral feeding
  The patient's body length will be measured on the electronic infant scale. Z-scores for weight for age (WAZ) was obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
The change of ostomy volume | From the the day starting the enteral nutrition to the fourth week.
  The amount of fistula form the ostomy bag will be recorded at the first day, the 14th day and the 28th day of the enteral nutrition.
Z-scores of head circumference | 4 weeks day after enteral feeding
  Z-scores were obtained from the World Health Organization Anthro software and WHO Child Growth Standards.
Cholestasis | 4 weeks day after enteral feeding
  The diagnostic criteria include the requirement of parenteral nutrition administration for a duration exceeding 2 weeks and an elevated direct bilirubin level > 34 mmol/L
The incidence rate of septicemia | Prior to complete enteral nutrition
  The impact of enteral nutrition (including enteral nutrition and breast milk) on the occurrence of septicemia in pediatric patients following enterostomy
The incidence rate of colitis | Prior to complete enteral nutrition
  The impact of enteral nutrition (including enteral nutrition and breast milk) on the occurrence of colitis in pediatric patients following enterostomy
D-lactic acid | One month after surgery
  Effect of enteral nutrition's impact on postoperative D-lactic acid level
D-lactic acid | Reaching full enteral feeding
  Effect of enteral nutrition's impact on postoperative D-lactic acid level
Adiponectin | One month after surgery
  Effect of enteral nutrition's impact on postoperative Adiponectin level
Adiponectin | Reaching full enteral feeding
  Effect of enteral nutrition's impact on postoperative Adiponectin level
leptin | One month after surgery
  Effect of enteral nutrition's impact on postoperative leptin level
leptin | Reaching full enteral feeding
  Effect of enteral nutrition's impact on postoperative leptin level
Overall duration of parenteral nutrition | 4 weeks day after enteral feeding
  For patients who cannot obtain sufficient nutrition through enteral feeding for more than 5 days, consideration should be given to providing parenteral nutrition support

CONTACTS AND LOCATIONS:
Overall Officials: Tian Qian, M.D., Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No